CLINICAL TRIAL: NCT01912105
Title: Evaluation of a Closed Suction System to Remove Secretions From the Endotracheal Tube: a Randomized Trial
Brief Title: Evaluation of a Closed Suction System to Remove Secretions From the Endotracheal Tube
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Principal Investigator, Antonio Pesenti, Prof., Azienda Ospedaliera San Gerardo di Monza
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 180-20130326
Record Dates: First submitted 2013-06-10; First posted 2013-07-30 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Intubation; Expected Duration of Ventilation > 48h
Keywords: endotracheal tube; ct scan; cleaning device; biofilm; mechanical ventilation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment (Experimental): Airway Medix Closed Suction System
  Interventions: Device: Airway medix closed suction system
- control (Active Comparator): standard closed suctioning systems
  Interventions: Device: standard closed suctioning systems

INTERVENTIONS:
Device: Airway medix closed suction system
  Arms: treatment
Device: standard closed suctioning systems
  Arms: control

SUMMARY:
Cleaning the endotracheal tube with a specifically designed device results in lower amount of secretions at extubation, assessed by micro CT scan

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted to an ICU
* 18 years old or more
* expected to be intubated for more than 48 hours
* less than 24 hours from intubation
* fraction of inspired oxygen set at the ventilator <80%

Exclusion Criteria:

* Current or past participation in another intervention trial conflicting with the present study
* expected survival less than 24 hours
* Acute severe asthma
* Use of Extracorporeal membrane oxygenation (ECMO) or candidates for ECMO
* Double lumen endotracheal tube in place
* Conditions which pose the patient at high risk if inadvertent endotracheal tube displacement occurs (laryngeal edema, cervical spine trauma, upper airways diseases with difficult reintubation)
* other contraindications posed by staff physicians

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-04; Primary Completion 2014-06 (Actual); Study Completion 2014-07 (Actual)

PRIMARY OUTCOMES:
Volume of secretions | within 12 hours after extubation
  Volume of secretions retained inside the endotracheal tube, assessed by micro ct scan

SECONDARY OUTCOMES:
adverse events | until extubation, death or tracheostomy (approximately 2 weeks)
  report of major and minor adverse events related to the use of the device

OTHER OUTCOMES:
endotracheal tube colonization | within 48 hours after extubation
  assessed by microbiologic testing of the endotracheal tube lavage fluid

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Pesenti, MD, Principal Investigator — San Gerardo Hospital; Giacomo Bellani, MD PhD, Study Director — San Gerardo Hospital
Locations (1):
- Azienda Ospedaliera San Gerardo, Monza, Italy

REFERENCES:
- [Background] Berra L, Coppadoro A, Bittner EA, Kolobow T, Laquerriere P, Pohlmann JR, Bramati S, Moss J, Pesenti A. A clinical assessment of the Mucus Shaver: a device to keep the endotracheal tube free from secretions. Crit Care Med. 2012 Jan;40(1):119-24. doi: 10.1097/CCM.0b013e31822e9fe3. PMID 21926595
- [Derived] Coppadoro A, Bellani G, Bronco A, Lucchini A, Bramati S, Zambelli V, Marcolin R, Pesenti A. The use of a novel cleaning closed suction system reduces the volume of secretions within the endotracheal tube as assessed by micro-computed tomography: a randomized clinical trial. Ann Intensive Care. 2015 Dec;5(1):57. doi: 10.1186/s13613-015-0101-9. Epub 2015 Dec 30. PMID 26714807